CLINICAL TRIAL: NCT00609141
Title: A Phase I Study of IMC-A12 (Anti-IGF-I Receptor Monoclonal Antibody, NSC #742460) in Children With Relapsed/Refractory Solid Tumors
Brief Title: IMC-A12 in Treating Young Patients With Relapsed or Refractory Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor or Other Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00363; NCI-2009-00363 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ADVL0712; CDR0000585700; ADVL0712 (Other: COG Phase I Consortium); ADVL0712 (Other: CTEP); U01CA097452 (NIH)
Record Dates: First submitted 2008-02-02; First posted 2008-02-06 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive, Peripheral | interventions — cixutumumab

ARMS (1):
- Treatment (monoclonal antibody therapy) (Experimental): Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 4 weeks for up to 2 years in the absence of unacceptable toxicity or disease progression.
  Interventions: Biological: cixutumumab; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: cixutumumab — Given IV
  Other Names: anti-IGF-1R recombinant monoclonal antibody IMC-A12; IMC-A12
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I clinical trial is studying the side effects and best dose of IMC-A12 in treating young patients with relapsed or refractory Ewing sarcoma/peripheral primitive neuroectodermal tumor or other solid tumors. Monoclonal antibodies, such as IMC-A12, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) or recommended phase II dose of IMC-A12 (cixutumumab) in children with relapsed or refractory solid tumors using a limited dose-escalation strategy.

II. To define and describe the toxicities of this drug in children with relapsed or refractory solid tumors.

III. To characterize the pharmacokinetics of this drug in children with relapsed or refractory solid tumors.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of this drug in children with relapsed or refractory solid tumors within the confines of a phase I study.

II. To obtain initial phase II efficacy data on the antitumor activity of this drug in children with Ewing sarcoma/peripheral primitive neuroectodermal tumor (PNET).

III. To examine change in IGF-IR and insulin receptor (IR) levels and IGF-IR and IR activation in lymphocytes as biomarkers of IMC-A12 action and specificity.

IV. To evaluate the effect of this drug on circulating levels of proteins involved in linear growth and glucose homeostasis, including IGF-I, IGF-II, IGF-BP3, growth hormone, insulin, and C-peptide.

V. To develop exploratory data concerning biomarkers of activity.

OUTLINE: This is a dose-escalation study.

Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 4 weeks for up to 2 years in the absence of unacceptable toxicity or disease progression.

Patients undergo blood sample collection periodically for pharmacokinetic, immunogenicity, and other correlative studies. Samples are analyzed for serum levels of IGF-I, IGF-II, IGF-BP3, growth hormone, insulin, and C-peptide; trough concentrations and PK sampling; and biomarkers, including IGF-IR expression and phosphorylation and insulin receptor expression and phosphorylation via immunoprecipitation and Western immunoblotting. Tumor tissue samples from patients with Ewing sarcoma/peripheral PNET are banked for future research.

After completion of study treatment, patients are followed at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor

  * Relapsed or refractory disease
  * No central nervous system (CNS) tumor or lymphoma
  * Histological confirmation may have been made at original diagnosis or at relapse
* Current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Measurable or evaluable disease
* Patients with Ewing sarcoma/peripheral primitive neuroectodermal tumor (PNET) must have tissue blocks or slides available

  * Study chair must be notified if tissue blocks or slides are not available
* Karnofsky performance status (PS) ≥ 50% (patients > 10 years of age) and Lansky (PS) ≥ 50% (patients ≤ 10 years of age)

  * Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Creatinine clearance or radioisotope GFR ≥ 70 mL/min OR serum creatinine based on age/gender as follows:

  * 1 to < 2 years (males and females 0.6 mg/dL)
  * 2 to < 6 years (males and females 0.8 mg/dL)
  * 6 to < 10 years (males and females 1.0 mg/dL)
  * 10 to < 13 years (males and females 1.2 mg/dL)
  * 13 to < 16 years (males 1.5 mg/dL and females 1.4 mg/dL)
  * ≥ 16 years (males 1.7 mg/dL and females 1.4 mg/dL)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN) for age
* SGPT (ALT) ≤ 110 μ/L (for the purpose of this study, the ULN for SGPT is 45 μ/L)
* Serum albumin ≥ 2 g/dL
* Patients with known bone marrow metastatic disease will be eligible for study but not evaluable for hematologic toxicity

  * Patients must not be known to be refractory to red cell or platelet transfusion
* Patients with solid tumors without bone marrow involvement must meet the following criteria:

  * Peripheral absolute neutrophil count ≥ 1,000/μL
  * Platelet count ≥ 100,000/μL (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment)
  * Hemoglobin ≥ 8.0 g/dL (may receive RBC transfusions)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* No uncontrolled infection
* No known type I or type II diabetes mellitus
* Able to comply with the safety monitoring requirements of the study, in the opinion of the investigator
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to IMC-A12
* Fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study
* At least 7 days since prior and no concurrent hematopoietic growth factors

  * Growth factors that support platelet or white cell number or function can only be administered for culture-proven bacteremia or invasive fungal infection
* At least 7 days since prior and no concurrent biologic antineoplastic agents
* At least 6 weeks since prior monoclonal antibodies
* At least 3 months since prior total body irradiation (TBI), craniospinal external radiotherapy (XRT), or ≥ 50% radiotherapy to the pelvis
* At least 2 weeks since prior local XRT (small port)
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* More than 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosourea)
* More than 7 days since prior and no concurrent systemic corticosteroids
* Prior stem cell transplant or rescue allowed provided there has been no evidence of active graft-versus-host-disease within the past 2 months
* No prior monoclonal antibody therapy targeting the IGF-IR
* No concurrent chemotherapy, radiotherapy, or immunotherapy
* No concurrent anticancer agents
* No concurrent insulin or growth hormone therapy
* No other concurrent investigational drugs

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Adverse events as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 | Weekly during each course
  Toxicity tables will be constructed to summarize the observed incidence by severity and type of toxicity.
MTD or recommended phase II dose | During course 1
  MTD will be the maximum dose at which fewer than one-third of patients experience dose-limiting toxicity (DLT). DLT is defined as any hematological and non-hematological toxicities that is possible, probably, or definitely attributed to IMC-A12.
Pharmacokinetics of IMC-A12 | At baseline, days 1, 8, 15, 22, and 28 of course 1, and days 15 and 28 of course 2

SECONDARY OUTCOMES:
Response rate (complete or partial response) in patients with Ewing sarcoma/peripheral PNET | Up to 30 days after completion of treatment
  Confidence intervals will be constructed according to the method of Chang and O'Brien to account for the two-stage design.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Malempati, Principal Investigator — COG Phase I Consortium
Locations (1):
- COG Phase I Consortium, Arcadia, California, United States